CLINICAL TRIAL: NCT06635317
Title: Efficacy of Arpirin in Preventing Venous Thromboembolism in Total Knee and Hip Replacement
Brief Title: Efficacy of Aspirin in Preventing Venous Thromboembolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Ana Luisa Galicia Zamalloa, MD, MSc, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 151.2022; 151.2022 (Other: ISSSTE)
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Venous Thromboembolism (VTE); Total Joint Arthroplasty; Total Hip Arthroplasty (THA)
Keywords: Aspirin; Venous thromboembolism; Total knee replacement; Total hip replacement; Thromboprophylaxis
MeSH Terms: conditions — Venous Thromboembolism | interventions — Aspirin; Enoxaparin

STUDY DESIGN:
Intervention Model Description: All patients who underwent a preoperative Doppler ultrasound of the lower extremities to screen for VTE and received antibiotic prophylaxis with cephalothin 1 gram intravenously.
  At six hours post-surgery, patients in the aspirin group received enoxaparin, 40 mg/day subcutaneously for 3 days, and aspirin, 100 mg/day orally for 25 days. Patients in the enoxaparin group received enoxaparin, 40 mg/day subcutaneously for 28 days, with the dose reduced to 20 mg for patients weighing less than 50 kg or with an estimated glomerular filtration rate less than 30 mL/min/1.73 m².
  Additionally, all patients received pneumatic compression stockings postoperatively for at least 21 days as standard care.
  Physical therapy was initiated on the day of surgery or postoperative day 1 and continued daily throughout the hospital stay.
  Postoperative wound care and Doppler ultrasound evaluations were performed at two and four weeks postoperatively to detect any evidence of VTE.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Long term aspirin group (Active Comparator): Long term aspirin group received enoxaparin, 40 mg/day subcutaneously for 3 days, and aspirin, 100 mg/day orally for 25 days
  Interventions: Drug: Aspirin
- Enoxaparin group (Active Comparator): enoxaparin group received enoxaparin, 40 mg/day subcutaneously for 28 days, with the dose reduced to 20 mg for patients weighing less than 50 kg or with an estimated glomerular filtration rate less than 30 mL/min/1.73 m².
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: Aspirin — 100 mg/day orally for 25 days
  Arms: Long term aspirin group
Drug: enoxaparin — 40 mg/day subcutaneously for 28 days, with the dose reduced to 20 mg for patients weighing less than 50 kg or with an estimated glomerular filtration rate less than 30 mL/min/1.73 m².
  Arms: Enoxaparin group

SUMMARY:
Efficacy of aspirin and enoxaparin in preventing venous tromboembolism was compared after total knee or hip arthroplasty.

DETAILED DESCRIPTION:
Background: Venous thromboembolism (VTE) remains a significant risk following joint replacements, despite advancements in prevention strategies. Aspirin-based therapies have gained popularity due to their perceived safety, ease of administration, and supportive evidence.This study aimed to compare the efficacy of aspirin and enoxaparin in preventing VTE after total knee or hip arthroplasty.

Methods: Sixty patients undergoing primary total knee or hip arthroplasty were randomized to receive either aspirin or enoxaparin. The primary outcome was symptomatic VTE within 90 days. Patients were followed up for Doppler ultrasound evaluations.

ELIGIBILITY:
Inclusion Criteria:

* All patients provided written informed consent.
* All patients who underwent primary total hip or total knee arthroplasty for osteoarthritis

Exclusion Criteria:

* preoperative anticoagulation (direct oral anticoagulant, warfarin, IMPROVE Bleeding Score more or equal to 7, dual antiplatelet therapy)
* medical contraindications (allergy, cancer, cardiac disease, kidney disease, or bleeding disorder precluding anticoagulation).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-24 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Symptomatic VTE | 90 days

SECONDARY OUTCOMES:
Wound bleeding | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- ISSSTEP, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No